CLINICAL TRIAL: NCT06760754
Title: Examining the Feasibility and Impact of a Clinic-based Food Farmacy and Digital Culinary Medicine Program Among Cancer Survivors Treated in a Safety Net Hospital
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1732; NCI-2024-10265 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Waitlist Control (Experimental): Participants will be assessed for study eligibility and randomized to study
  Interventions: Dietary Supplement: Digital culinary medicine intervention
- Intervention Group (Experimental): Participants will be assessed for study eligibility and randomized to study
  Interventions: Dietary Supplement: Digital culinary medicine intervention

INTERVENTIONS:
Dietary Supplement: Digital culinary medicine intervention — Participants will receive 30lbs of healthy foods through an on-site hospital-base food pantry

SUMMARY:
The goal of this study is to develop and test the feasibility of a theory-driven digital culinary medicine program among food insecure cancer survivors referred from the University of Texas MD Anderson Cancer Center Oncology Clinic at LBJ to the LBJ Food Farmacy program.

DETAILED DESCRIPTION:
Primary Objective:

Determine the feasibility of study recruitment goal, intervention adherence rate, attrition rate, data completion rate, and program satisfaction rate.

Secondary Objective:

Assess the preliminary efficacy of the digital culinary medicine intervention to improve diet quality, food security, quality of life, and downstream biological indicators of cardiometabolic health from baseline to post-intervention, as well as from baseline to 6 month follow up, among food insecure cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivors treated at the MD Anderson Oncology Program at LBJ Hospital over 18 years of age.
* Screen positive for food insecurity using the 2 question clinic-screener (Hunger Vital Signs)
* Receive referral to the LBJ Food Farmacy.
* Are within the first 5 years off of acute cancer treatment.
* Self-report having internet access.
* Self-report as being able to speak and read English or Spanish.
* Willing to complete study assessments.

Exclusion Criteria:

* Unwilling or unable to complete study assessments
* Anyone under 18 years of age
* Self-report to not speak or read English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Raber, DRPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org